CLINICAL TRIAL: NCT05798247
Title: Cutaneous Diphtheria in France : an Observational, Retrospective Study of Epidemiological, Clinical, Microbiological and Therapeutic Characteristics
Brief Title: Cutaneous Diphtheria in France : Observational, Retrospective Study of Patient Characteristics
Acronym: OEDIPE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Centre d'Epidémiologie et de Santé Publique des Armées (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-CHITS-013
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Corynebacterium Diphtheriae Infection
Keywords: Cutaneous; Diphteria
MeSH Terms: conditions — Diphtheria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cutaneous diphteria: The study group consists of all the patients suffering from cutaneous diphtheria in metropolitan France and for which microbiological data were registered by the National Reference Center fo corynebacteria of the diphteriae complex between 2018 and 2022.
  Interventions: Other: Characteristics description

INTERVENTIONS:
Other: Characteristics description — Caregivers who follow the patients of the study group will be contacted to collect these patients clinical and epidemiological characteristics

SUMMARY:
Toxigenic cutaneous diphtheria is a notifiable disease that is re-emerging in the world and particularly in France. A better description of the epidemiological characteristics, as well as a refinement of the clinical characteristics of patients with cutaneous diphtheria, are essential to better understand this pathology, which has important public health issues and whose diagnosis absence can have catastrophic consequences for the patient and their contacts. Microbiological data (species identification, toxigenicity or not, resistance profile...) will be transmitted by the national reference center for corynebacteria of the diphtheriae complex and then caregivers who have managed the corresponding patients with cutaneous diphtheria will be contacted.

ELIGIBILITY:
Inclusion Criteria:

* Culture or PCR positive skin samples for corynebacteria diphtheria, ulcerans, pseudotuberculosis, belfantii or rouxii
* Patient living in metropolitan France

Exclusion Criteria:

- Patient opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population corresponds to all metropolitan French patients suffering from cutaneous diphtheria for which microbiological data were registered between 2018 and 2022 by the National Reference Center for corynebacteria of the diphteriae complex.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Patients epidemiological data description | 3 months
  Epidemiological data will be collected to describe the studied population (age, sex, place of birth, vaccination status...)
Patients clinical data description | 3 months
  Clinical data will be collected to describe the studied population (history, description of lesions, disease evolution, complications...)
Patients microbiological data description | 3 months
  Microbiological data will be collected to describe the studied population (species identification, toxigenicity, presence of a co-infection...)
Patients therapeutic data description | 3 months
  Therapeutic data will be collected to describe the studied population (antibiotic therapy, duration of treatment, search for an eradication a posteriori...)

SECONDARY OUTCOMES:
Comparison of antibiotic therapy duration to national recommendations issued by the High Committee of Public Health | 3 months
  Duration of antibiotic therapy implemented by clinicians will be compared to national recommendations
Comparison of immunization status monitoring to national recommendations issued by the High Committee of Public Health | 3 months
  Monitoring of immunization status or not will be collected
Comparison of patient post infection vaccination status to national recommendations issued by the High Committee of Public Health | 3 months
  Post-infection vaccination or not will be collected
Comparison of patient microbiological follow-up to national recommendations issued by the High Committee of Public Health | 3 months
  Microbiological follow-up with eradication research or not will be collected.
Comparison of post-infection serological sampling to national recommendations issued by the High Committee of Public Health | 3 months
  Whether a post-infection serological sampling was performed or not will be collected.
Comparison of patient isolation procedures to national recommendations issued by the High Committee of Public Health | 3 months
  Patient isolation or not will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien DUTASTA, MD, Study Director — SSA
Locations (42):
- France (42):
  - Institut Hospitalo-Universitaire de Marseille, Marseille, Bouches-du-Rhône
  - CHU de Dijon, Dijon, Bourgogne-Franche-Comté
  - CHU de Caen, Caen, Calvados
  - Centre Hospitalier de Brive, Brive-la-Gaillarde, Corrèze
  - Centre Hospitalier de Guingamp, Pabu, Côtes d'Armor
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes, Essonne
  - CHU Bordeaux, Bordeaux, Gironde
  - Hôpital Louis Pasteur (HCC), Colmar, Haut-Rhin
  - Centre Hospitalier Alpes-Leman CHAL, Contamine-sur-Arve, Haute-Savoie
  - Centre Hospitalier de Briançon, Briançon, Hautes-Alpes
  - Centre Hospitalier de Lourdes, Lourdes, Hautes-Pyrénées
  - Hôpital Ambroise Paré (AP-HP), Boulogne-Billancourt, Hauts-de-Seine
  - Hôpital Américain de Paris, Neuilly-sur-Seine, Hauts-de-Seine
  - CHU de Montpellier, Montpellier, Hérault
  - CHRU de Tours, Chambray-lès-Tours, Indre-et-Loire
  - Groupement Hospitalier Nord Dauphiné, Bourgoin, Isère
  - CHU de Nantes, Nantes, Loire-Atlantique
  - Centre Hospitalier Régional d'Orléans, Orléans, Loiret
  - Centre Hospitalier de Cahors, Cahors, Lot
  - Centre Hospitalier Cholet, Cholet, Maine-et-Loire
  - Centre Hospitalier de Saint-Lo, Saint-Lô, Manche
  - CHU de Lille, Lille, Nord
  - Centre Hospitalier de Valenciennes, Valenciennes, Nord
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez, Pays de la Loire Region
  - Centre d'endocrinologie, Cabestany, Pyrénées Orientales
  - Hôpital Edouard Herriot (HCL), Lyon, Rhône
  - Hôpital Croix rousse (HCL), Lyon, Rhône
  - Centre Hospitalier William Morey, Chalon-sur-Saône, Saône-et-Loire
  - Centre Hospitalier de Mâcon, Mâcon, Saône-et-Loire
  - Hôpital Avicenne Bobigny (AP-HP), Bobigny, Seine-Saint-Denis
  - CHU d'Amiens, Amiens, Somme
  - Hôpital Nord Franche-Comté, Trévenans, Territoire De Belfort
  - Hôpital Henri Mondor (AP-HP), Créteil, Val-de-Marne
  - HIA Sainte Anne, Toulon, VAR
  - Centre Hospitalier d'Avignon, Avignon, Vaucluse
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon, Vendée
  - Hôpital Saint Joseph, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital La Pitié Salpêtrière, Paris
  - Groupement Hospitalier Diaconesses Croix Saint Simon, Paris
  - CHU de Toulouse - Hôpital La Grave, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernard KA, Pacheco AL, Burdz T, Wiebe D. Increase in detection of Corynebacterium diphtheriae in Canada: 2006-2019. Can Commun Dis Rep. 2019 Nov 7;45(11):296-301. doi: 10.14745/ccdr.v45i11a04. eCollection 2019 Nov 7. PMID 31755876
- [Background] Martini H, Soetens O, Litt D, Fry NK, Detemmerman L, Wybo I, Desombere I, Efstratiou A, Pierard D. Diphtheria in Belgium: 2010-2017. J Med Microbiol. 2019 Oct;68(10):1517-1525. doi: 10.1099/jmm.0.001039. PMID 31418673
- [Background] Jaton L, Kritikos A, Bodenmann P, Greub G, Merz L. [European migrant crisis and reemergence of infections in Switzerland]. Rev Med Suisse. 2016 Apr 13;12(514):749-53. French. PMID 27263151
- [Background] Morgado-Carrasco D, Riquelme-Mc Loughlin C, Fusta-Novell X, Fernandez-Pittol MJ, Bosch J, Mascaro JM Jr. Cutaneous Diphtheria Mimicking Pyoderma Gangrenosum. JAMA Dermatol. 2018 Feb 1;154(2):227-228. doi: 10.1001/jamadermatol.2017.4786. No abstract available. PMID 29282460
- [Background] Pandit N, Yeshwanth M. Cutaneous diphtheria in a child. Int J Dermatol. 1999 Apr;38(4):298-9. doi: 10.1046/j.1365-4362.1999.00658.x. No abstract available. PMID 10321948
- [Background] Wagner KS, White JM, Lucenko I, Mercer D, Crowcroft NS, Neal S, Efstratiou A; Diphtheria Surveillance Network. Diphtheria in the postepidemic period, Europe, 2000-2009. Emerg Infect Dis. 2012 Feb;18(2):217-25. doi: 10.3201/eid1802.110987. PMID 22304732
- [Background] Gower CM, Scobie A, Fry NK, Litt DJ, Cameron JC, Chand MA, Brown CS, Collins S, White JM, Ramsay ME, Amirthalingam G. The changing epidemiology of diphtheria in the United Kingdom, 2009 to 2017. Euro Surveill. 2020 Mar;25(11):1900462. doi: 10.2807/1560-7917.ES.2020.25.11.1900462. PMID 32209165
- [Background] Koopman JS, Campbell J. The role of cutaneous diphtheria infections in a diphtheria epidemic. J Infect Dis. 1975 Mar;131(3):239-44. doi: 10.1093/infdis/131.3.239. PMID 805182
- [Background] de Benoist AC, White JM, Efstratiou A, Kelly C, Mann G, Nazareth B, Irish CJ, Kumar D, Crowcroft NS. Imported cutaneous diphtheria, United Kingdom. Emerg Infect Dis. 2004 Mar;10(3):511-3. doi: 10.3201/eid1003.030524. PMID 15109425
- [Result] Chene L, Morand JJ, Badell E, Toubiana J, Janvier F, Marthinet H, Suppini JP, Valois A, Texier G, Brisse S, Dutasta F OEDIPE Study Group. Cutaneous diphtheria from 2018 to 2022: an observational, retrospective study of epidemiological, microbiological, clinical, and therapeutic characteristics in metropolitan France. Emerg Microbes Infect. 2024 Dec;13(1):2408324. doi: 10.1080/22221751.2024.2408324. Epub 2024 Sep 30. PMID 39324172
- See also: Related Info — https://www.santepubliquefrance.fr/maladies-et-traumatismes/maladies-a-prevention-vaccinale/diphterie/documents/rapport-synthese/enquete-nationale-de-couverture-vaccinale-france-janvier-2011.-couverture-vaccinale-contre-la-grippe-saisonniere-dans-les-groupes-cibles-et-mesur
- See also: Related Info — https://www.ecdc.europa.eu/sites/default/files/media/en/publications/Publications/Diphtheria-cutaneous-EU-July-2015.pdf